CLINICAL TRIAL: NCT05595486
Title: Baby2Home (B2H) Mobile Health Application: A Randomized-Controlled Trial
Brief Title: Baby2Home (B2H) Mobile Health Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Northwestern University (Other)
Responsible Party: Principal Investigator, Emily Miller, Associate Professor, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STU00216659; 1R01HD105499-01 (NIH)
Record Dates: First submitted 2022-05-05; First posted 2022-10-27 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: COVID-19 Pandemic; Health Knowledge, Attitudes, Practice; Perinatal Depression; Mental Health Wellness; Post Partum Depression
MeSH Terms: conditions — COVID-19; Behavior; Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Families will be randomized into either the control or intervention group.
Who Masked: Outcomes Assessor
Masking Description: The research team abstracting the data and performing the analyses will be masked to the randomization arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): As a pragmatic trial, usual care will be defined by contemporary clinical standards. For maternal care, this includes a comprehensive medical visit between 4-12 weeks postpartum. This visit includes utilization of a validated screen for postpartum depression and, if that screen is positive, a clinical assessment and initiation of treatment (e.g. pharmacotherapy or referral for psychotherapy). In addition, this visit includes a discussion of contraception as well as supportive education on breastfeeding. For paternal care, clinical standards are gleaned from the AAP, ACOG, and USPSTF reports outlining mental health screening, reproductive health, and vaccine uptake. For infant care, standard pediatric care from the AAP and Bright Futures periodicity timeline and guidelines will be used. In addition, assignment in this arm will be given surveys at baseline, 1M, 2M, 4M, 6M, and 12M.
- Baby2Home Intervention (Experimental): Families randomized to the intervention arm will receive the B2H services. B2H is a novel digitized CC-based intervention delivered via a smartphone app available on iOS or Android phones, built by combining two successful programs: NICU2Home+ app and CC services. Using the UCD methodologies, AI-based communication within the app will include education for mothers and fathers on the standard of care regarding self-care and newborn care after hospital discharge as well as education, reminders and scheduling for recommended preventative healthcare services for themselves and their new infant.
  Interventions: Other: Baby2Home Mobile Application

INTERVENTIONS:
Other: Baby2Home Mobile Application — Baby2Home is a digital health intervention designed to bridge the resultant gaps in obstetrics and pediatrics healthcare services for new families over the first year of life.
  Arms: Baby2Home Intervention

SUMMARY:
The COVID-19 pandemic has transformed healthcare delivery; arguably, the fields of obstetrics and pediatrics have experienced some of the greatest changes as they have transitioned away from their role as a medical home and into more of an urgent care model of care. Baby2Home is a digital health intervention designed to bridge the resultant gaps in obstetrics and pediatrics healthcare services for new families over the first year of life. This randomized controlled trial will evaluate whether, compared to usual care, Baby2Home 1) improves maternal, paternal, and infant health service utilization outcomes over the first year postpartum, 2) improves maternal and paternal patient reported outcomes, and 3) reduces racial/ethnic and income-based disparities in preventive health services utilization and parental patient reported outcomes.

DETAILED DESCRIPTION:
The transition to new parenthood is marked by dramatic changes in social roles and responsibilities. To support new parents, obstetric and pediatric healthcare surrounding this transition is designed with a supportive focus to facilitate new parents' navigation of the attendant life changes. The COVID-19 pandemic has altered healthcare delivery in ways that have limited these supportive obstetrics and pediatric services provided at the beginning of new parenthood. Consequently, aspects of preventative healthcare, such as monitoring for symptoms of postpartum depression, discussing optimal birth control options, educating parents on recommended adult and pediatric vaccinations, and providing anticipatory guidance on infant wellness, are less robust. In addition, without professional guidance and support, outcomes of foundational importance to new parents, such as perceived stress, depressive and anxiety symptoms, or parenting and breast-feeding self-efficacy, are worse. Moreover, the COVID-19 pandemic has underscored the impact of the social determinants of health on new family wellness, with racial/ethnic minority and low-income families being differentially impacted by COVID-19 pandemic driven healthcare delivery changes. Recognizing the potential for longitudinal changes in healthcare delivery engendered by the COVID-19 pandemic, a scalable, patient-centered, equity-focused intervention designed to bridge gaps in healthcare services around the transition to new parenthood is needed.

"Bridging gaps in healthcare delivery to COVID-19 for parent and infants from birth through the first year of life" aims to evaluate Baby2Home (B2H) a patient-informed digital healthcare intervention that s is specifically responsive to the COVID-19 pandemic's impact on new families, with a focus on health equity for racial/ethnic minority and low-income families. B2H builds upon previous digital health successes while incorporating the evidence-based collaborative care model for mental health support. B2H is designed to mitigate the adverse effects of healthcare delivery changes in response to the COVID-19 pandemic and to improve health for mothers, fathers, and infants over the first year of life. Developed from feedback given by new parents who delivered during the COVID-19 pandemic, B2H provides 1) parental education about their own physical and mental health, 2) infant wellness resources and tracking of recommended healthcare services, 3) parental mental health screening and support, and 4) systematic case review to optimize the health of new families. The investigators will test the efficacy of B2H via a randomized control trial. In total, 640 diverse families will be randomly to either usual care or B2H intervention arm to evaluate whether, compared to usual care, B2H health services utilization and patient reported outcomes of foundational important to new families. addition, the investigators will evaluate the impact of B2H on racial/ethnic and income-based disparities observed in both services utilization and patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Delivery at Prentice Women's Hospital or Women and Infants Hospital of Rhode Island
* Viable term infant (≥ 37 weeks)
* First live born child
* English speaking
* Age 18 years old or greater
* Access to a smartphone
* Access to a working email address

Exclusion Criteria:

* No smartphone access
* Infant death
* Infant requires NICU admission
* Known severe mental illness of either parent (e.g., bipolar disorder, schizophrenia)
* SARS-CoV-2 infection without clinical clearance
* History of IPV (intimate partner violence) with current partner (would exclude partner)
* Concurrent enrollment in studies that may affect the outcome of the trial (or vice versa)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 642 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Completion of preventive health services utilization for all family members (birthing, non-birthing, and infant) | Baseline through 1 year postpartum
  The primary outcome defined as positive if all of the items below are met for all family members:
  1. optimal maternal preventive health services utilization over the 1st year postpartum (including attendance at the comprehensive postpartum visit, receives chosen contraceptive method, and undergoes postpartum depression screening)
  2. optimal paternal/co-parental preventive health services utilization over the 1st year postpartum (including receiving recommended vaccinations for new parents, if desires a male-driven contraceptive option, receives chosen method, and undergoes screening for depression)
  3. optimal infant preventive health services utilization over the 1st year postpartum (including attending all AAP recommended wellness visits, receiving all AAP recommended vaccines, and receiving breast milk for 6 months of life)

SECONDARY OUTCOMES:
Number of participants who attend comprehensive postpartum visit (birthing parent) | At least once between 4 and 12 weeks postpartum
  Subject returns for a comprehensive medical care at least once between 4 and 12 weeks postpartum. This visit should include documented elements of physical health, mood, mode of infant feeding, contraception, preventive health, and any comorbidities.
Completion of postpartum depression screening (birthing parent) | Through study completion, up to 12 months
  Subject completes a validated screen for postpartum depression and, if the screen is positive, receives a recommendation for treatment. To assess depressive symptoms, birthing will take the 9-item Patient Health Questionnaire (PHQ). This is scored on a Likert-type scale from 0 - 3 (Not at all to Nearly everyday). A lower score reflects minimal depression and a higher score reflects severe depression.
Number of participants who received contraception (birthing and non-birthing parent) | Through study completion, up to 12 months
  If a subject desires a contraceptive method, they receives chosen method. Receipt of contraception can be an actual insertion of device (implant or IUD), receipt of injection, receipt of sterilization (BTL or vasectomy, if vasectomy is confirmed to have been performed), or prescription for a combined hormonal contraceptive method.
Number of participants who received the recommended vaccinations (non-birthing parent) | Through study completion, up to 12 months
  Subject receives influenza and TDaP vaccines before 12 months postpartum.
Completion of postnatal depression screening for non-birthing parent | Through study completion, up to 12 months
  Subject completes a validated screen for depression. To assess depressive symptoms, non-birthing parents will take the 9-item Patient Health Questionnaire (PHQ). This is scored on a Likert-type scale from 0 - 3 (Not at all to Nearly everyday). A lower score reflects minimal depression and a higher score reflects severe depression.
Number of participants who attended well-child visits for the infant | Through study completion, up to 12 months
  Subject attends all AAP recommended wellness visits. Attendance at each visit will be derived from both patient-report (via B2H) and through ROIs from the pediatrician offices. Preference will be given to the ROIs, but if this not available, patient-report will be used as equal. If these data points are conflicting, patient-report will supersede the medical record.
Number of participants who received the recommended vaccinations for infant | Through study completion, up to 12 months
  Subject receives all AAP recommended vaccinations. This information will be ascertained from the ROIs from the pediatrician offices. Recognizing various vaccine schedules, this will be determined as a binary variable at 12 months postpartum (and the % of vaccines received).
Continued breastfeeding for infants until 6 months | Through study completion, up to 6 months
  This outcome will be patient-reported. The investigators will evaluate this outcome as positive if breastmilk is a source of nutrition until 6 months.
  The primary analysis will be of all subjects who were eligible for breastfeeding (i.e., excluding those unable to breastfeed due to a medical complication). Investigators will perform secondary analyses in which individuals who do not desire breastfeeding and did not initiate breastfeeding will not be considered in this component of outcomes.
Duration of breastfeeding (birthing parent) | Through study completion, up to 6 months
  This outcome will be patient-reported. The investigators will also evaluate as an ordinal outcome of total duration (months) of any breastfeeding and total duration (months) of exclusive breastfeeding.
  The primary analysis will be of all subjects who were eligible for breastfeeding (i.e., excluding those unable to breastfeed), but the investigators will perform secondary analyses in which individuals who do not desire breastfeeding and did not initiate breastfeeding will not be considered in this component of outcomes.
Patient reported outcomes: stress symptoms (for birthing and non-birthing parent) | Month 1, 2, 4, 6, and 12
  To assess stress, birthing and non-birthing parents will take the 10-item Perceived Stress Scale (PSS). This is scored on a Likert-type scale from 0 - 4 (Never to Very often). Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Patient reported outcomes: depressive symptoms (for birthing and non-birthing parent) | Month 1, 2, 4, 6, and 12
  To assess depressive symptoms, birthing and non-birthing parents will take the 9-item Patient Health Questionnaire (PHQ). This is scored on a Likert-type scale from 0 - 3 (Not at all to Nearly everyday). A lower score reflects minimal depression and a higher score reflects severe depression.
Patient reported outcomes: anxiety symptoms (for birthing and non-birthing parent) | Month 1, 2, 4, 6, and 12
  To assess anxiety, birthing and non-birthing parents will take the 7-item Generalized Anxiety Disorder Scale. This is scored on a Likert-type scale from 0 - 3 (Not at all to Nearly everyday). A lower score reflects minimal anxiety and a higher score reflects severe anxiety.
Patient reported outcomes: global health status (for birthing and non-birthing parent) | Month 1, 2, 4, 6, and 12
  To assess health status, birthing and non-birthing parents will take the 10-item PROMIS Global Health Scale. This is scored on a Likert-type scale from 5 - 1 (Excellent to Poor). A higher score indicates better health status.
Patient reported outcomes: relationship assessment (for birthing and non-birthing parent) | Month 1, 2, 4, 6, and 12
  To assess relationship status, birthing and non-birthing parents will take the 14-item Revised Dyadic Adjustment Scale (RDAS). This is scored on a Likert-type scale from 0 - 5 (Everyday to Never). Scores on the RDAS range from 0 to 69 with higher scores indicating greater relationship satisfaction and lower scores indicating greater relationship distress. The cut-off score for the RDAS is 48 such that scores of 48 and above indicate non-distress and scores of 47 and below indicate marital/relationship distress.
Patient reported outcomes: self-efficacy (for birthing and non-birthing parent) | Month 1, 2, 4, 6, and 12
  To assess self-efficacy, birthing and non-birthing parents will take the 10-item PROMIS Self-Efficacy Scale. This is scored on a Likert-type scale from 1 - 5 (I am not at all confident to I am very confident). A higher score indicates a higher sense of general self-efficacy.
Patient reported outcomes: parenting self-efficacy (for birthing and non-birthing parent) | Month 12
  To assess parenting self-efficacy, birthing and non-birthing parents will take the 17-item Parenting Sense of Competence Scale. This is scored on a Likert-type scale from 1 - 6 (Strongly Disagree to Strongly Agree). A higher score indicates a higher parenting sense of competency.
Patient reported outcomes: breastfeeding self-efficacy (for birthing parent) | Month 1, 2, 4, 6, and 12
  To assess breastfeeding self-efficacy, birthing parents will take the 12-item Breastfeeding Self-Efficacy scale. This is scored on a Likert-type scale from 1 - 7 (Strongly Disagree to Strongly Agree). A higher score indicates a better/more positive outcome towards breastfeeding.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Craig, MD, Study Director — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (2):
- United States (2):
  - Northwestern Medicine Prentice Women's Hospital, Chicago, Illinois
  - Women and Infant's Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang E, Lewkowitz AK, Unger JA, Garfield CF, Miller ES. Smartphone Applications to Support Perinatal Mental Health. Obstet Gynecol. 2026 Feb 1;147(2):229-238. doi: 10.1097/AOG.0000000000006139. Epub 2025 Dec 18. PMID 41411652